CLINICAL TRIAL: NCT04504487
Title: "Early Versus Routine Drain Removal After Live Liver Donor Hepatectomy- a Randomized Controlled, Open Label, Pilot Study".
Brief Title: Early Versus Routine Drain Removal After Live Liver Donor Hepatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ILBS/LIVEDONORS/01
Record Dates: First submitted 2020-07-30; First posted 2020-08-07 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-01

CONDITIONS: Liver Transplant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early drain removal - POD3 (Experimental): Drain removal on POD3 if drain bilirubin is less than 3mg/dl and serous in nature.
  Interventions: Other: Drain Removal
- Routine Drain Removal (Placebo Comparator): Drain removed routinely when the output is less than 100ml and serous in nature
  Interventions: Other: Drain Removal

INTERVENTIONS:
Other: Drain Removal — Abdominal drain placed during surgery removal

SUMMARY:
It's a randomized control trial to compare early drain removal versus standard drain removal after donor hepatectomy in terms of donor outcomes. We will analyse the data and elucidate the safety of early drain removal using 3x3 rule with routine drain removal.

DETAILED DESCRIPTION:
* Prophylactic abdominal drainage after donor right hepatectomy for LDLT has been a common or even mandatory practice in most transplant centres.
* This serves to monitor the occurrence of postoperative intraabdominal bleeding and is used for the detection and drainage of any bile leakage.
* Below table mentions both advantages and disadvantages of prophylactic drain placement after hepatectomy.

Advantages

1. Early detection of haemorrhage
2. Early detection of bile leak
3. Early reintervention Disadvantages

1. Increased rates of intraabdominal and wound infection, 2. Increased abdominal pain, 3. Decreased pulmonary function, 4. Prolonged hospital stay, 5. Bowel injury.

* Our study in ILBS for ALF donors, the overall complication rate was 20% as per Clavien-Dindo classification, of which a majority (15.9%) had grade 1 or 2 complications. Major complications (3b and above) were seen in 4 (1.0%) patients. Biliary complications were noted in 1.7% only.
* In a study by Japanese group concluded that 3 × 3 rule is clinically feasible and allows for the early removal of the drain tube with minimum infection risk after liver resection. The ''3 x 3 rule'': the drain will be removed when the drain fluid bilirubin concentration is <3 mg/dl on day 3 after operation.
* In our institute we remove drain routinely, when output is less than 100ml and serous. That is usually on postoperative day 5-7.
* There is no randomized control trail done in donor hepatectomy comparing early versus standard drain removal.

ELIGIBILITY:
Inclusion Criteria:

* • Donors evaluated as per institutional protocol for donor hepatectomy and found fit

  * Those who consent

Exclusion Criteria:

* Patients refusing to consent for inclusion in the study.
* Left lateral hepatectomy.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2021-01-28 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2022-02-25 (Actual)

PRIMARY OUTCOMES:
safety of drain removal using 3x3 rule - overall complications. | patient will be followed upto 3 months after surgery
  Comprehensive complication index (CCI) - clavin dindo classification

SECONDARY OUTCOMES:
Post operative pain relief | patient will be followed upto 3 months after surgery
  using Visual analogue score
Bile leak | patient will be followed upto 3 months after surgery
  standard ISGLS definition - drain bilirubin measured in mg/dl.
Length of hospital stay | patient will be followed upto 3 months after surgery
  calculated from the day of admission to day of discharge, and based on the number of nights spent in hospital
Surgical Site Infection (SSI) | patient will be followed upto 3 months after surgery
  patient has at least one of the following:
  1. purulent drainage from the superficial incision.
  2. organism(s) identified from an aseptically-obtained specimen from the superficial incision or subcutaneous tissue by a culture or non-culture based microbiologic testing method which is performed for purposes of clinical diagnosis or treatment (for example, not Active Surveillance Culture/Testing (ASC/AST)).
  3. superficial incision that is deliberately opened by a surgeon, physician* or physician designee and culture or non-culture based testing of the superficial incision or subcutaneous tissue is not performed AND patient has at least one of the following signs or symptoms: localized pain or tenderness; localized swelling; erythema; or heat.
  4. diagnosis of a superficial incisional SSI by a physician* or physician designee.
reintervention rate | patient will be followed upto 3 months after surgery
  defined as any additional abdominal intervention ( surgical or radiological) during the same hospital stay after the primary operation
readmission rate | patient will be followed upto 3 months after surgery
  90 day readmission rate - any hospital admission after the index admission.

CONTACTS AND LOCATIONS:
Locations (1):
- ILBS - Parthiban, Delhi, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Durairaj P, Pamecha V, Mohapatra N, Patil NS, Sindwani G. Early drain removal after live liver donor hepatectomy is safe - a randomized controlled pilot study. Langenbecks Arch Surg. 2023 Sep 5;408(1):350. doi: 10.1007/s00423-023-03088-9. PMID 37670194
- See also: Prospective Validation of Optimal Drain Management "The 3 × 3 Rule" after Liver Resection — https://pubmed.ncbi.nlm.nih.gov/27138885/
- See also: Living Donor Liver Transplantation for Acute Liver Failure: Donor Safety and Recipient Outcome — https://pubmed.ncbi.nlm.nih.gov/30861306/
- See also: Criteria for drain removal following liver resection — https://pubmed.ncbi.nlm.nih.gov/23027077/